CLINICAL TRIAL: NCT07157930
Title: Relationship Between Prenatal Hormonal Markers in Young Adults With Joint Hypermobility: The Role of the 2D:4D Digit Ratio
Brief Title: Prenatal Hormonal Markers and Sleep Characteristics in Young Adults With Joint Hypermobility
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Nigde Omer Halisdemir University
Other Study IDs: Joint Hypermobility and 2D:4D
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Joint Hypermobility; Healty Controls; Sleep; Androgen Effect; Hormonal
Keywords: joint hypermobility; sleep; 2D:4D; digit ratios
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young Adults With Joint Hypermobility: Joint hypermobility makes individuals more vulnerable to trauma through increased joint range of motion, changes in neuromuscular reflexes, and decreased joint position sense. The Beighton Scoring system is widely used to distinguish individuals with generalized joint hypermobility from those without.In adults up to 50 years of age, a score of ≥5 out of 9 indicates hypermobility, while in adults over 50, a score of ≥4 out of 9 is considered positive for hypermobility.
  The study will include young adults aged 18-35 with joint hypermobility. It has been reported in the literature that estrogen may be associated with connective tissue laxity and joint hypermobility. The 2D:4D digit ratio will be assessed and compared with young adults without joint hypermobility.
  Interventions: Behavioral: The Beighton Scoring system; Behavioral: 2D:4D Digit Ratio
- Healthy Controls (without joint hypermobility): This group consisted of individuals without generalized joint hypermobility, confirmed by a Beighton score below the diagnostic cut-off. This study will include young adults aged 18-35 who do not have joint hypermobility.The Beighton Scoring system is widely used to distinguish individuals with generalized joint hypermobility from those without.In adults up to 50 years of age, a score of ≥5 out of 9 indicates hypermobility, while in adults over 50, a score of ≥4 out of 9 is considered positive for hypermobility. Individuals with musculoskeletal, neurological, or systemic conditions that may affect joint mobility will be excluded from the study.
  Interventions: Behavioral: The Beighton Scoring system; Behavioral: 2D:4D Digit Ratio

INTERVENTIONS:
Behavioral: The Beighton Scoring system — The Beighton Scoring System is widely used to distinguish individuals with generalized joint hypermobility from those without. The Beighton Scoring System consists of: • Passive dorsiflexion of the fifth metacarpophalangeal joint • Passive hyperextension of the elbow • Passive hyperextension of the knee joint • Passive placement of the thumb on the flexor side of the forearm • Forward flexion of the trunk In adults up to 50 years of age, a score of ≥5 out of 9 indicates joint hypermobility, while in adults over 50, a score of ≥4 out of 9 is considered positive for joint hypermobility.
Behavioral: 2D:4D Digit Ratio — The lengths of the second (2D) and fourth (4D) digits will be measured separately on both hands. Measurements will be taken with the participants' hands placed on a flat surface with the palms facing upward. Digit length will be defined as the distance from the midpoint of the proximal crease at the base of the finger to the distal tip of the finger. A digital caliper with a precision of 0.01 mm will be used, and two separate measurements will be obtained for each finger, with the mean value recorded. Based on these measurements, the 2D:4D digit ratio will be calculated for each hand by dividing the length of the second digit by that of the fourth digit. To enhance reliability, assessments will be performed independently by two different researchers, and inter-rater agreement will be evaluated.

SUMMARY:
Joint hypermobility is a clinical condition characterized by joints having a range of motion beyond their normal limits. Hormonal factors are thought to play a role in the development of joint hypermobility. One of the most significant indicators of prenatal androgen exposure is considered the ratio of the lengths of the second and fourth fingers (2D:4D). The 2D:4D digit ratio refers to the ratio of the lengths of the second finger (2D; index digit ) and the fourth finger (4D; ring digit). Evidence suggests that the 2D:4D ratio is developmentally stable and stabilizes from the second trimester of pregnancy onward.

To our knowledge, intrauterine androgen exposure (2D:4D) has not been examined in populations with joint hypermobility.

Therefore, the planned study aimed to examine the 2D:4D digit ratio in young adults with joint hypermobility and compare it with that of individuals without joint hypermobility.

DETAILED DESCRIPTION:
Estrogen affects collagen metabolism and connective tissue structure, which can lead to increased ligament laxity at high levels. Increased estrogen and progesterone during pregnancy cause significant loosening of connective tissue, which can contribute to temporary joint hypermobility. Physiological conditions such as pregnancy and menopause can cause hormonal changes, increasing the risk of joint hypermobility through fluid retention and connective tissue changes.

Testosterone, on the other hand, is a hormone that strengthens muscle mass and tendon structure, while at low levels it can cause connective tissue to remain looser. Therefore, the combination of high estrogen and relatively low testosterone, particularly in women of reproductive age, may contribute to the higher prevalence of hypermobility.

Therefore, the aim of the planned study was to examine the 2D:4D digit ratio in young adults with joint hypermobility and compare this ratio with individuals without joint hypermobility.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-35
* Individuals who scored 5 out of 9 or higher on the Beighton score
* Control group: Those with a Beighton score of ≤ 4

Exclusion Criteria:

* Individuals with any pathology related to the musculoskeletal system
* Individuals diagnosed with metabolic, neurological, or genetic diseases (tissue diseases such as Ehlers-Danlos syndrome and Marfan syndrome)
* Those with a history of surgery within the last 6 months
* Those who are pregnant or breastfeeding

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study planned to include individuals with (Beighton skorlamasına göre 9 üzerinden 5 ve daha fazla puan alan) and without joint hypermobility. Individuals between the ages of 18 and 35 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Beighton Scoring System | 1 month
  Individuals will be assessed for joint hypermobility (Beighton Scoring System) by a physical therapist. The Beighton Scoring System is widely used to distinguish individuals with generalized joint hypermobility from those without. The Beighton Scoring System consists of:
  * Passive dorsiflexion of the fifth metacarpophalangeal joint
  * Passive hyperextension of the elbow
  * Passive hyperextension of the knee joint
  * Passive placement of the thumb on the flexor side of the forearm
  * Forward flexion of the trunk In adults up to 50 years of age, a score of ≥5 out of 9 indicates joint hypermobility, while in adults over 50, a score of ≥4 out of 9 is considered positive for joint hypermobility.
2D:4D Digit Ratio | 1 month
  The lengths of the second (2D) and fourth (4D) digits will be measured separately on both hands. Measurements will be taken with the participants' hands placed on a flat surface with the palms facing upward. Digit length will be defined as the distance from the midpoint of the proximal crease at the base of the finger to the distal tip of the finger. A digital caliper with a precision of 0.01 mm will be used, and two separate measurements will be obtained for each finger, with the mean value recorded. Based on these measurements, the 2D:4D digit ratio will be calculated for each hand by dividing the length of the second digit by that of the fourth digit. To enhance reliability, assessments will be performed independently by two different researchers, and inter-rater agreement will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fink B, Manning JT, Neave N. The 2nd-4th digit ratio (2D:4D) and neck circumference: implications for risk factors in coronary heart disease. Int J Obes (Lond). 2006 Apr;30(4):711-4. doi: 10.1038/sj.ijo.0803154. PMID 16261185
- [Result] Engelbert RH, Bank RA, Sakkers RJ, Helders PJ, Beemer FA, Uiterwaal CS. Pediatric generalized joint hypermobility with and without musculoskeletal complaints: a localized or systemic disorder? Pediatrics. 2003 Mar;111(3):e248-54. doi: 10.1542/peds.111.3.e248. PMID 12612280
- [Result] Smits-Engelsman B, Klerks M, Kirby A. Beighton score: a valid measure for generalized hypermobility in children. J Pediatr. 2011 Jan;158(1):119-23, 123.e1-4. doi: 10.1016/j.jpeds.2010.07.021. Epub 2010 Sep 17. PMID 20850761
- [Result] Gruber PC, Fuller LC. Lipoatrophy semicircularis induced by trauma. Clin Exp Dermatol. 2001 May;26(3):269-71. doi: 10.1046/j.1365-2230.2001.00812.x. PMID 11422172